CLINICAL TRIAL: NCT02143440
Title: The Initial Assessment of Daily Insulin Dose in Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012273
Record Dates: First submitted 2014-05-17; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes.
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Newly diagnosed type 2 patients (Other): The initial assessment of daily insulin dose.
  Interventions: Behavioral: The initial assessment of daily insulin dose.

INTERVENTIONS:
Behavioral: The initial assessment of daily insulin dose.

SUMMARY:
To investigate the daily dose of insulin in newly diagnosed Chinese type 2 diabetic patients who use the continuous subcutaneous insulin infusion (CSII) as the initial therapy.

ELIGIBILITY:
Inclusion Criteria:

All participants with type 2 diabetes, diagnosed by World Health Organization criteria, were recruited from outpatient of the Endocrinology Department in Shanghai Renji Hospital.

Exclusion Criteria:

Patients who had a history of coronary heart disease, abnormal renal function, active liver disease, chronic metabolic acidosis (including diabetic ketoacidosis), or severe chronic gastrointestinal disease.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
When the glucose level decreased to about 10 mmol/L | 72-96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China